CLINICAL TRIAL: NCT01260428
Title: Arterial Oxygenation During Hypoxia : Effects of an Added Expiratory Resistance
Brief Title: Effects of Expiratory Pressure on Arterial Oxygenation During Hypoxia
Acronym: hypex
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AGIR à Dom (Other)
Responsible Party: Sponsor
Other Study IDs: 10-AGIR-2
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Hypoxia
Keywords: hypoxia; O2 diffusion and convection; cardiac output; PEEP; Effects of hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy active subjects: with and without high altitude intolerance
  Interventions: Device: threshold PEEP

INTERVENTIONS:
Device: threshold PEEP — Various set of pressures : 0, 5, 10 cm H20; pursed lips breathing

SUMMARY:
Altitude tolerance correlates with the level of oxygenation achieved. The aim of the present study is to investigate whether increased expiratory pressure within the thorax is able to improve oxygenation during hypoxic hypoxia.

DETAILED DESCRIPTION:
Two types of procedures will be tested in a random order, interspaced by resting periods : threshold PEEP set at 5,10 and 15 cm of water and pursed leap breathing.

Subjects will be tested at rest, and during light exercise (30% of sea level predicted VO2max).

FiO2 will be set at 12.5% (4000 m). fc, VE, PETCO2, TA, ECG, cardiac output, and tissular oxygenation will be monitored.

ELIGIBILITY:
Inclusion Criteria :

* active (> 2 hrs/week physical activity)
* adult
* non smoking volunteers

Exclusion Criteria :

* cardiac, respiratory, neuromuscular, metabolic pathology

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample with mounteneering experience
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-02

PRIMARY OUTCOMES:
SpO2 | mean over 1 minute
  after three minutes of PEEP vs spontaneous breathing

SECONDARY OUTCOMES:
peripheral HbO2/DeoxyHb | 1 min
  after three minutes of PEEP / PLB vs. spontaneous breathing
cardiac output | mean over 1 min
  after three min of PEEP vs. spontaneous breathing
pattern of breathing (fR, VT, PETCO2) | 1 min
  after three min of PEEP vs. spontaneous breathing

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Wuyam, MD, PhD, Principal Investigator — University Hospital, Grenoble; Samuel Vergès, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Hugo NESPOULET, MsC, Study Chair — Université Joseph Fourier
Locations (1):
- CHU de Grenoble, La Tronche, Isere, France